CLINICAL TRIAL: NCT03398343
Title: Nutritional Therapy on Underweight Critically Ill Patients: an Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Mirela Jobim de Azevedo, Professor, Hospital de Clinicas de Porto Alegre
Other Study IDs: CAAE 45677715.2.0000.5327
Record Dates: First submitted 2016-03-15; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2017-02

CONDITIONS: Underweight; Critical Illness
MeSH Terms: conditions — Thinness; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Critically ill patients with body mass index (BMI) inferior to 20 kg/m2 have worse outcomes compared to normal and overweight patients. The impact nutrition therapy in this population is not yet stablished. There is a concern that too low caloric intake might worse their malnutrition; on the other hand, overfeeding is always a risk with serious consequences.

The hypothesis of this study is that nutritional support, especially caloric and protein intake, can influence the outcome of underweight critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Ages eligible for study: 18 years and older
* Gender eligible: both
* Nutrition therapy: enteral, parenteral feeding, nothing by mouth

Exclusion Criteria:

* Palliative care
* Exclusively oral nutrition
* Pregnancy
* Life expectancy inferior 24 hours
* ICU readmission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with body mass index (BMI) inferior to 20 kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | through study completion (up to a year)
  All patients will be followed until live hospital discharge or death

SECONDARY OUTCOMES:
ICU length of stay | through study completion (up to a year)
  patients will be followed until ICU discharge or death
Need and duration of mechanical ventilation | through study completion (up to a year)
  all patients for which mechanical ventilation is necessary will be followed until it is no longer necessary

CONTACTS AND LOCATIONS:
Locations (1):
- HCPA, Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Viana MV, Gross LA, Tavares AL, Tonietto TA, Costa VL, Moraes RB, Azevedo MJ, Viana LV. Functional assessment and mortality in underweight critically ill patients one year after hospital discharge: A prospective cohort study. Clin Nutr ESPEN. 2023 Jun;55:151-156. doi: 10.1016/j.clnesp.2023.03.007. Epub 2023 Mar 15. PMID 37202039
- [Derived] Viana MV, Tavares AL, Gross LA, Tonietto TA, Costa VL, Moraes RB, Azevedo MJ, Viana LV. Nutritional therapy and outcomes in underweight critically ill patients. Clin Nutr. 2020 Mar;39(3):935-941. doi: 10.1016/j.clnu.2019.03.038. Epub 2019 Apr 5. PMID 31003789